CLINICAL TRIAL: NCT05289024
Title: Pragmatic Implementation of Mindful Awareness in Body Oriented Therapy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Kathryn A. Hansen, Medical Director, Vanderbilt University Medical Center
Other Study IDs: 201931
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Non-pharmacologic Management of Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MABT utilizers: Chronic pain patients receiving MABT in an interdisciplinary clinic as part of their standard of care.
  Interventions: Behavioral: Mindful Awareness in Body-Oriented Therapy

INTERVENTIONS:
Behavioral: Mindful Awareness in Body-Oriented Therapy — Up to 8 individually delivered clinical sessions

SUMMARY:
This is a one group study using a hybrid implementation design.

DETAILED DESCRIPTION:
The proposed pilot study will collect preliminary data to support a larger hybrid effectiveness-implementation study designed to examine the implementation of the evidence-based Mindful Awareness in Body-oriented Therapy (MABT), delivered by massage therapists, on patient and implementation science outcomes in an interdisciplinary chronic pain clinic. The combined foci of this mixed-methods pilot study is expected to provide an indication of implementation success, highlight implementation processes, and show treatment effectiveness on health outcomes.1 MABT is a mind-body therapy designed to teach interoceptive awareness skills for symptom management and emotion regulation. The proposed pilot study uses mixed methods and a single-group repeated measures design to explore MABT implementation and to estimate the effect of MABT to reduce symptomatic distress in the treatment of chronic pain at the Osher Center for Integrative Medicine at Vanderbilt Clinic (OCIM).

ELIGIBILITY:
Inclusion Criteria:

* Patient attending clinic and who received a referral to MABT

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients attending an integrative health center
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of referrals to MABT | 24 months
  Total number of referrals from clinicians within the clinic to MABT
Total number of MABT visits | 24 months
  Total number of MABT visits utilized during study period
Number of referrals to MABT from a Psychologist | 24 months
  Count of how many of the total referrals came from Psychologists
Number of referrals to MABT from a Nurse Practitioner | 24 months
  Count of how many of the total referrals came from Nurse Practitioners
Number of referrals to MABT from a Physical Therapist | 24 months
  Count of how many of the total referrals came from Physical Therapists
Number of referrals to MABT from a Massage Therapist | 24 months
  Count of how many of the total referrals came from Massage Therapists

SECONDARY OUTCOMES:
Health related quality of life | 32 weeks
  PROMIS-29 This 29 question survey contains 7 domains each captured by 4 questions using a 5 point Likert scale with 0 being the least and 5 representing the most of each concept. the 29th question is an 11 point pain scale with 0 being no pain and 10 being the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen KA, Abu-Rish Blakeney E, Price CJ. Implementation Outcomes From a Pilot Study of Mindful Awareness in Body-Oriented Therapy (MABT) as a Chronic Pain Treatment Modality in an Integrative Health Clinic. Glob Adv Integr Med Health. 2025 Feb 7;14:27536130251319244. doi: 10.1177/27536130251319244. eCollection 2025 Jan-Dec. PMID 39925451